CLINICAL TRIAL: NCT06180902
Title: Comparing Fluid Responsiveness Assessment Methods in Patients With Impaired Consciousness: A Comprehensive Crossover Study Examination
Brief Title: Comparing Fluid Responsiveness Assessment Methods in Patients With Impaired Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology (Other)
Responsible Party: Principal Investigator, Valery Likhvantsev, Principal Investigator, Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPASS
Record Dates: First submitted 2023-12-11; First posted 2023-12-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypotension; Cognitive Impairment
Keywords: Hypotension; Cognitive Impairment; Fluid Responsiveness; Intensive Care; Fluid Infusion
MeSH Terms: conditions — Hypotension; Cognitive Dysfunction | interventions — Central Venous Pressure

STUDY DESIGN:
Intervention Model Description: For all patients included in the study, a designated algorithm will be applied. The initial phase of the clinical study, aimed at evaluating responsiveness to infusion therapy, starts with a precise measurement of the inferior vena cava's diameter. After a brief two-minute interval subsequent to the measurement, the focus shifts to the assessment of central venous pressure. A further two-minute pause following the central venous pressure evaluation signals the commencement of the passive leg raise test, an essential element in the protocol. The conclusion of the passive leg raise test is followed by a fifteen-minute waiting period, which precedes the start of the fluid challenge, completing the thorough evaluation sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluid responsiveness testing (Experimental): In our clinical study to evaluate infusion therapy responsiveness, we'll start by measuring the inferior vena cava diameter. Two minutes later, we'll assess central venous pressure. After another two-minute pause, the passive leg raise test begins, followed by a 15-minute wait. Then, we conduct the fluid challenge. Post-evaluation, we administer balanced crystalloid solutions at 1000 ml, infused at 15 ml/kg/h, adjusting for any previous infusions during the fluid challenge.
  Interventions: Diagnostic Test: Inferior vena cava's diameter ratio; Diagnostic Test: Central venous pressure; Diagnostic Test: Passive leg raising test; Diagnostic Test: Fluid challenge; Procedure: Fluid infusion

INTERVENTIONS:
Diagnostic Test: Inferior vena cava's diameter ratio — In mechanical ventilation, the Inferior Vena Cava's maximum diameter (IVCmax) is measured at peak inspiration, and minimum diameter (IVCmin) at expiration's end. The Distensibility Index (IVCDI) is calculated as [(IVCmax - IVCmin) / IVCmin] × 100%. In spontaneous breathing, IVCmax is the diameter at expiration's end, and IVCmin at inspiration's end. The Collapse Index (IVCCI) is [(IVCmax - IVCmin) / IVCmax] × 100%.
  Clinically, an IVCDI/IVCCI ≥ 18% indicates a 'responder'. Values < 18% denote 'non-responders'.
Diagnostic Test: Central venous pressure — In our protocol, patients lie flat, connected to a saline-filled system for intravenous infusion via a central venous catheter. The system, starting from the subclavian catheter, extends to the 2nd to 3rd intercostal space at the mid-axillary line. The tube's end is raised perpendicular to the bed until saline flow stops, marking the liquid level. The height from the mid-axillary line to this point is measured in millimeters. If the liquid column falls below the mid-axillary line, indicating continuous flow, the CVP is negative, and the catheter is closed to block air entry. CVP readings are taken at exhalation's end.
  CVP interpretation:
  * CVP ≤ 12 mmHg (16.3 cm H2O) indicates a responder.
  * CVP > 12 mmHg (16.3 cm H2O) indicates a non-responder.
Diagnostic Test: Passive leg raising test — In our protocol, the patient starts flat for initial CVP measurement. Then, the bed is tilted to 45 degrees for the first measurements: Systolic/Diastolic Blood Pressure, Mean Arterial Pressure, and Pulse Pressure (Systolic - Diastolic). Next, the bed is adjusted to elevate the feet, creating a 135-degree angle between torso and legs. After 90 seconds, the second set of measurements, including CVP, is taken. The patient is then returned to the initial position.
  Interpreting results:
  A responder is indicated by:
  * Over 10% Pulse Pressure (PP) increase in the second measurement;
  * The ratio of PP change to CVP change (∆PP / ∆CVP) > 1;
  * Second measurement CVP ≤ 12 mmHg (16.3 cm H2O).
  A non-responder is indicated by the presence at least one of the following:
  * Less than 10% PP increase in the second measurement;
  * The ratio of PP change to CVP change (∆PP / ∆CVP) ≤ 1;
  * Second measurement CVP > 12 mmHg (16.3 cm H2O).
  Other Names: PLR-test
Diagnostic Test: Fluid challenge — In our clinical procedure, patients start horizontally for initial measurements: Systolic, Diastolic, Mean Arterial, Pulse Blood Pressures, and Central Venous Pressure (CVP). Then, they receive a balanced crystalloid solution at 4 ml/kg body weight at maximum permissible infusion rate. After infusion, a second measurement set identical to the first is taken.
  Interpretation:
  A responder is indicated by:
  * Pulse Pressure (PP) increase > 10% in second measurement;
  * Ratio of PP change to CVP change (∆PP / ∆CVP) > 1;
  * Second CVP measurement ≤ 12 mmHg (16.3 cm H2O).
  A non-responder is indicated by the presence at least one of the following:
  * PP increase < 10% in second measurement;
  * Ratio of PP change to CVP change (∆PP / ∆CVP) ≤ 1;
  * Second CVP measurement > 12 mmHg (16.3 cm H2O).
  Other Names: FC
Procedure: Fluid infusion — After assessing infusion therapy responsiveness, patients receive balanced crystalloid solutions at 1000 ml, infused at 15 ml/kg/hour, accounting for any prior infusions. Effectiveness evaluation follows, involving cardiac output reassessment (initially measured upon study enrollment). Effectiveness is determined by a ≥10% increase in cardiac output in the second measurement compared to the first. This is quantified as: [(CO(after) - CO(before)) / CO(before)] × 100% ≥ 10%, where CO(after) is the post-infusion cardiac output and CO(before) the pre-infusion output.

SUMMARY:
Hypotension is a significant precursor to unfavorable clinical outcomes. To determine whether infusion therapy can positively impact the management of hypotension, several evaluative tests can be utilized. These include assessing the collapsibility and distensibility indices of the inferior vena cava, conducting a passive leg raising (PLR) test, and performing a fluid challenge (FC).

Technologically advanced methods leveraging dynamic testing are capable of real-time prediction of a patient's response to infusion therapy. Nonetheless, the use of systolic pressure variability (SPV), pulse pressure variability (PPV), and stroke volume variability (SVV) is often limited by the prohibitive costs of the necessary equipment. In contrast, the PLR test and FC are not subject to this limitation.

Despite being deemed unreliable by numerous clinical protocols, static measurements of central venous pressure (CVP) or pulmonary capillary wedge pressure (PCWP) persist in usage among certain traditionalists within the medical community. It must be noted that the patient's baseline state and the unique clinical context are pivotal in determining the precision of these methodologies. For example, the PLR test may yield limited information in fully conscious patients, and the prognostic value of CVP measurements is significantly diminished in cases of pneumothorax and hydrothorax.

Regrettably, there is a paucity of data on the prognostic utility of these tests in patients with altered levels of consciousness, despite their growing presence in intensive care units. This gap underscores the necessity for comprehensive studies that evaluate the predictive efficacy of infusion therapy responsiveness in patients with concurrent hypotension and impaired consciousness.

Purpose of the study: to investigate the sensitivity and specificity of methods for assessing fluid responsiveness in patients with hypotension and decreased level of consciousness.

DETAILED DESCRIPTION:
Hypotension often precedes adverse clinical outcomes, prompting an investigation into the efficacy of infusion therapy in its management. The study employs a variety of tests for assessment, including evaluation of the inferior vena cava's collapsibility and distensibility indices, passive leg raise (PLR) tests, and fluid challenge (FC) procedures.

Dynamic testing methods, including systolic pressure variability (SPV), pulse pressure variability (PPV), and stroke volume variability (SVV), offer predictions of real-time responses to infusion therapy. However, the high costs of the necessary equipment restrict widespread application. In contrast, passive leg raise (PLR) and fluid challenge (FC) tests are more accessible due to lower costs.

Despite skepticism in various clinical protocols regarding reliability, traditional measures such as central venous pressure (CVP) and pulmonary capillary wedge pressure (PCWP) continue to be favored in certain medical circles. Considering the patient's baseline condition and specific clinical context is critical when applying such methods. For instance, the PLR test may be less informative in fully conscious patients, and the value of CVP measurements decreases in cases like pneumothorax and hydrothorax.

A notable deficiency exists in data concerning the prognostic value of tests in patients with altered consciousness levels, a scenario frequently encountered in intensive care settings. This situation underscores the urgent need for comprehensive research into the predictive accuracy of infusion therapy response in patients who have coexisting hypotension and impaired consciousness.

The study aims to examine the sensitivity and specificity of fluid responsiveness assessment methods in hypotensive patients with reduced consciousness. The protocol begins by measuring the diameter of the inferior vena cava, followed by an evaluation of central venous pressure. After a brief interval, the passive leg raise (PLR) test is performed, succeeded by a 15-minute waiting period. Subsequently, an infusion load test is carried out. Next, a balanced crystalloid solution of 1000 ml at a rate of 15 ml/kg/h is administered, taking into account any previous infusions during the fluid challenge.

In the study, adherence to the intention-to-treat principle is planned for all analyses. Data distribution will be assessed using the Kolmogorov-Smirnov test with Lilliefors correction or the Shapiro-Wilk test. Descriptive data will be presented as percentages, means ± SD for normally distributed variables, or medians ± interquartile ranges for non-normally distributed variables. Qualitative characteristics will be reported as frequencies. P-values and confidence intervals will be provided for all comparative outcomes between two groups. All statistical tests will be two-tailed, with a significance threshold set at p < 0.05.

Outcomes for all binary variables, including primary and secondary outcomes, will be compared using the Chi-square test or Fisher's exact test, accounting for stratification variables. Comparative intergroup analysis of quantitative variables will be based on the Mann-Whitney U test or Student's t-test, depending on data distribution characteristics. Baseline data will include diagnostic test results such as true positives, true negatives, false positives, and false negatives. Diagnostic accuracy will be assessed using Area Under the Receiver Operating Characteristic curve (AUROC) and Area Under the Precision-Recall curve (AUPC). AUROC comparisons will be made using the DeLong method, with the optimal cutoff in ROC analysis determined according to Youden's index. Sensitivity, specificity, and predictive values of positive and negative results will also be evaluated. Cohen's Kappa will be used to assess test consistency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Hospitalization in an intensive care unit
* Level of consciousness on the FOUR scale ≤ 12 points
* Planned infusion therapy
* Presence of a central venous catheter or direct indication for catheterization
* The decision of the medical council to include the patient in the study

Exclusion Criteria:

* Pulmonary edema
* Absence of one or both lower extremities
* Chronic kidney disease according to KDIGO classification ≥ stage 3b
* Acute kidney injury grade 3
* Documented or suspected increased intracranial pressure (cerebral edema, brain compression, hydrocephalus, etc.).
* Presence of mitral valve regurgitation > grade 1
* Presence of aortic valve regurgitation > grade 1
* Patients previously enrolled in the "COMPASS" study in the period of 12 preceding hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of methods for assessing fluid responsiveness | Through study completion, an average of 1 year
  Sensitivity - proportion of actual positives that are correctly identified by the test.
  Specificity - proportion of actual negatives that are correctly identified by the test.

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, PhD, Principal Investigator — Federal Research and Clinical Center of Intensive Care Medicine and Rehabilitology
Locations (1):
- Federal Research and Clinical Center of Intensive Care Medicine and Rehabilitology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No